CLINICAL TRIAL: NCT00876941
Title: Efficacy/Effectiveness of Unhealthy Drug Use Screening/Brief Intervention Models
Brief Title: Assessing Screening Plus Brief Intervention's Resulting Efficacy (ASPIRE) to Stop Drug Use
Acronym: ASPIRE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Boston University (Other); RTI International (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DESPR DA025068; R01DA025068 (NIH); Grant Number: 1R01DA025068
Record Dates: First submitted 2009-04-06; First posted 2009-04-07 (Estimated); Last update posted 2014-10-02 (Estimated); Status verified 2012-02

CONDITIONS: Drug Usage; Drug Abuse; Drug Dependence
Keywords: Drug; Drug Use; Screening; Brief Intervention; Primary Care; Utilization
MeSH Terms: conditions — Substance-Related Disorders; Patient Acceptance of Health Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Standard Brief Intervention (Experimental)
  Interventions: Behavioral: Standard Brief Intervention
- Enhanced Brief Intervention (Experimental)
  Interventions: Behavioral: Enhanced Brief Intervention
- Control (Active Comparator)
  Interventions: Behavioral: Control: Information and Feedback

INTERVENTIONS:
Behavioral: Standard Brief Intervention — Intervention: Structured, brief negotiated interview.
  Intervention preparation and content: Preparation: review of ASSIST results; Content: The intervention involves 4 major parts: 1) establishing rapport and asking the subject for permission to raise the topic of drug use; 2) exploring the pros and cons of use; 3) providing feedback and assessing readiness to change; and 4) advising and negotiating a plan.
  Counselor: Health Promotion Advocate, High School graduate or GED minimum Training specific to the brief intervention: Didactic and experiential; competency demonstrated by observation and/or video recordings which are content scored using a standardized form.
  Contacts, Duration: One, 10-15 minutes.
  Communication content delivered to primary care physician: Results of screening and BI.
  Supervision: Weekly 1-hour meeting with supervisor to discuss job performance and discuss cases; biannual shadowing by supervisor.
  Other Names: BI-S
  Arms: Standard Brief Intervention
Behavioral: Enhanced Brief Intervention — Intervention: Less structured, motivational interview.
  Intervention preparation and content: Preparation: review of ASSIST, drug consequences (SIP-D), risk behaviors, CIDI Short Form, and medical record for discussion; Content: Motivational interviewing discussing above.
  Counselor: Master's level/Doctoral student.
  Training specific to the brief intervention: Didactic and experiential, followed by additional work towards, and confirmation of, proficiency using audio recordings coded for motivational interviewing content.
  Contacts, Duration: One plus offer of one optional booster contact, each 30-45 minutes; 2nd by telephone or in person depending on subject's preference; availability of counselor for further readiness discussions.
  Communication content delivered to primary care physician: Results of screening, BI, and plan including follow-up.
  Supervision: Weekly 1.5-hour meeting with supervisor with review of coded audio recordings.
  Other Names: BI-E
  Arms: Enhanced Brief Intervention
Behavioral: Control: Information and Feedback — Subjects randomized to the control group will not receive a BI at enrollment. But, all study subjects will receive screening and its results as part of the informed consent process (that they are at least at risk for drug use health hazards) along with a written list of resources available, including local options.
  Arms: Control

SUMMARY:
The objective of this study is to test whether screening and brief intervention for drug use among primary care patients leads to improved drug-related outcomes (such as decreased drug use and consequences).

DETAILED DESCRIPTION:
The efficacy of screening and brief intervention (SBI) for drug use among primary care patients is unknown. National organizations do not recommend universal screening. But policy is at odds with the evidence: federal efforts to disseminate SBI are underway, and reimbursement codes to compensate clinicians have been developed. Thus there is a need to study SBI for drug use. The objective of this study is to determine the efficacy of two models of brief intervention (BI) for decreasing drug use and consequences in primary care patients. In collaboration with a state project implementing SBI as part of a federal program, we will screen patients in a large hospital-based primary care practice for drug use. We will then enroll screen-positive subjects, randomly assign them to 1 of 3 groups, and follow them for 6 months. Subjects in 1 intervention group will be assigned to a standard BI model, conducted by trained health advocates implementing a Federal program locally. In another group, subjects will be assigned to an enhanced BI model that includes an optional booster contact and is conducted by master's-level counselors trained and monitored intensively. The control group will receive information (i.e., a written list of local resources to help people using drugs) and, at the end of six months, standard BI if they are still using drugs.

All subjects will be assessed regarding substance use and consequences, HIV risk behaviors, costs, healthcare utilization and receipt of substance dependence treatment. The primary outcome is drug use at 6 months; secondary outcomes are drug use consequences, including HIV risk behaviors, and receipt of substance dependence treatment (among those with dependence). We hypothesize that the standard BI and the enhanced BI will each have greater efficacy than screening and resource information alone for decreasing drug use, decreasing drug use consequences and HIV risk behaviors and increasing receipt of treatment for those with dependence.

Additionally, costs will also be compared. Results of this study re: efficacy and costs of brief intervention for drug use will be essential for making decisions about disseminating drug use SBI in primary care settings.

This study will enroll two cohorts:

1. We will enroll 450 subjects with an ASSIST Substance-Specific Involvement (SSI) Score of 4 or greater in order to test our primary hypotheses. Primary analyses (i.e., effect of each BI on unhealthy drug use) will be restricted to subjects with an ASSIST SSI Score of 4 or greater.
2. We will enroll an additional 200 subjects with an ASSIST SSI Score of 2 or 3, indicating some, but lower risk drug use. Patients with these scores are included in clinical interventions, but because there are no data on effectiveness in the literature, this cohort will not be included in primary analyses and instead will be included only in secondary and exploratory analyses. We will examine potential preventive effects of BI (either) on subjects with lower level drug use.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Arrived for a visit in primary care
* ASSIST Substance Specific Involvement Score of greater than or equal to 4 for subjects included in primary analyses; ASSIST Substance-Specific Involvement Scores of 2 or 3 for subjects included only in exploratory analyses
* No previous MASBIRT intervention in the past 3 months
* Fluent in English or Spanish
* Two contacts who can assist with locating the subject for follow-up
* Able to return to Boston Medical Center in the next 6 months for research study visits
* Not pregnant (because care systems and resources differ greatly for such subjects)
* Able to be interviewed by trained research staff (excluding those in acute discomfort or with significantly impaired cognition)

Exclusion Criteria:

* NOT 18 years of age or older
* NOT Arrived for a visit in primary care
* NO ASSIST Substance Specific Involvement Score of greater than or equal to 4 for subjects included in primary analyses; or NO ASSIST Substance-Specific Involvement Scores of 2 or 3 for subjects included only in exploratory analyses
* ANY previous MASBIRT intervention in the past 3 months
* NOT Fluent in English or Spanish
* FEWER THAN two contacts who can assist with locating the subject for follow-up
* NOT able to return to Boston Medical Center in the next 6 months for research study visits
* Pregnant (because care systems and resources differ greatly for such subjects)
* UN-Able to be interviewed by trained research staff (excluding those in acute discomfort or with significantly impaired cognition)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 589 (Actual)
Dates: Start 2009-04; Primary Completion 2012-10 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Drug use | Six Months

SECONDARY OUTCOMES:
Drug use consequences | Six Months
HIV risk behaviors | Six Months
Substance abuse treatment utilization | Six Months
Costs | Six Months

CONTACTS AND LOCATIONS:
Overall Officials: Richard Saitz, MD, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Alford DP, German JS, Samet JH, Cheng DM, Lloyd-Travaglini CA, Saitz R. Primary Care Patients with Drug Use Report Chronic Pain and Self-Medicate with Alcohol and Other Drugs. J Gen Intern Med. 2016 May;31(5):486-91. doi: 10.1007/s11606-016-3586-5. Epub 2016 Jan 25. PMID 26809204
- [Derived] Saitz R, Palfai TP, Cheng DM, Alford DP, Bernstein JA, Lloyd-Travaglini CA, Meli SM, Chaisson CE, Samet JH. Screening and brief intervention for drug use in primary care: the ASPIRE randomized clinical trial. JAMA. 2014 Aug 6;312(5):502-13. doi: 10.1001/jama.2014.7862. PMID 25096690